CLINICAL TRIAL: NCT06434350
Title: Enfortumab Vedotin With Radiation for Locally Advanced Bladder Cancer (CONSOLIDATE)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0071; NCI-2024-04592 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Bladder Cancer
MeSH Terms: interventions — enfortumab vedotin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enfortumab Vedotin with Radiation (Experimental): Particpants will receive enfortumab vedotin by vein over about 1-2 hours on Days 1 and 8 of every 28-day cycle. Two dose levels of enfortumab vedotin will be tested. The dose of enfortumab vedotin participants receive will depend on when the participant join the study.
  Participants will also receive radiation therapy 5 times a week (Monday through Friday) for about 4-5 weeks.
  Interventions: Drug: Enfortumab Vedotin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Enfortumab Vedotin — Given by IV
Radiation: Radiation Therapy — Given by Radiation Therapy

SUMMARY:
To learn if the combination of enfortumab vedotin plus radiation therapy could help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives:

1. Primary Objective #1: To estimate progression free survival for concurrent enfortumab vedotin with RT in locally advanced MIBC
2. Primary Objective #2: To evaluate the safety/tolerability of enfortumab vedotin with RT in participants with locally advanced MIBC
3. Primary Objective #3: To evaluate global health-related quality of life (HRQOL) using EQ-5D-5L, EORTC MIBC module, and EPIC bowel domain surveys

Secondary Objectives:

1. Secondary Objective #1: To estimate the overall survival at 12 months after study enrollment.
2. Secondary Objective #2: To estimate the metastasis free survival at 12 months after study enrollment.
3. Secondary Objective #3: To determine the treatment related toxicities associated with enfortumab vedotin with RT as part of definitive local therapy for advanced MIBC.
4. Secondary Objective #4: To estimate the freedom from GU events after enfortumab vedotin with RT
5. Exploratory Objective #1: To determine the association of translational biomarkers including peripheral blood tumor markers and urine tumor markers with participant outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of urothelial carcinoma of the bladder including patients with T4N0 and T1-4N2-3 disease. Participants with mixed urothelial carcinoma of bladder will also be included.
2. Be ≥ 18 years of age on the day of signing informed consent.
3. ECOG performance status 0-2. NOTE: If participants is unable to walk due to paralysis, but is mobile in a wheelchair, participants is ambulatory for the purpose of assessing their performance status.
4. The participant has the following baseline laboratory data:

   1. Hemoglobin ≥ 9 g/dL
   2. Platelet count ≥ 100 x 109 g/dL
   3. Creatinine clearance (CrCl) ≥ 30 mL/min as estimated per institutional standards (glomerular filtration rate [GFR] can also be used instead of CrCl)
   4. Absolute neutrophil count (ANC) ≥ 1500/mm3
5. Male participants must consistently use highly effective methods of birth control starting at screening and continue throughout study period and for at least 6 months after radiation completion
6. Female participants must consistently use highly effective methods of birth control starting at screening and continue throughout the study period and for at least 6 months after radiation completion As the CORe system in MDACC is set up as a one-step enrollment process, the above inclusion criteria will be assessed prior to CORe enrollment. Following CORe enrollment, the below inclusion criteria will be assessed.

1. Candidate for definitive local therapy to active disease per the discretion of the treating physicians.

Exclusion Criteria:

1. Has a diagnosis of active scleroderma, lupus, ulcerative colitis, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe radiation therapy.
2. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial as determined by the treating physician and/or member of the study team.
3. Distant metastatic disease beyond lymph node metastases, which by the discretion of the treating physician cannot be treated definitively in a radiation field
4. Has history of prior pelvic radiation therapy
5. Has ongoing clinically significant toxicity (Grade 2 or higher with exception of alopecia) associated with prior systemic therapy
6. History of uncontrolled diabetes mellitus within 3 months of enrollment. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥ 8% or HbA1c between 7 and < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
7. Has estimated life expectancy of less than 12 weeks
8. Has preexisting sensory or motor neuropathy Grade ≥ 2
9. Participants receiving ongoing systemic intravenous antimicrobial treatment for active infection at time of randomization
10. Participants have a known history of hepatitis B (defined as HBsAg reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. No testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
11. Has a known history of human immunodeficiency virus (HIV) infection. Testing is not required unless mandated by the local health authority.
12. Has conditions requiring high doses of steroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded. Inhaled or topical steroids are permitted in the absence of active autoimmune disease. Physiologic replacement doses of corticosteroids are permitted for participants with adrenal insufficiency.
13. Has a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
14. Has received a prior allogeneic stem cell or solid organ transplant.
15. Has active tuberculosis As the CORe system in MDACC is set up as a one-step enrollment process, the above inclusion criteria will be assessed prior to CORe enrollment. Following CORe enrollment, the below exclusion criteria will be assessed.

1. Is pregnant or expecting to conceive within the projected duration of the trial at the screening visit.

* Female participants of childbearing potential should have a negative urine or serum pregnancy within 6 weeks prior to study registration up to the first fraction of radiation.
* Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-09-24 (Estimated); Study Completion 2027-09-24 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Comron Hassanzadeh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org